CLINICAL TRIAL: NCT03268538
Title: Evaluation of Finger Wearable Device to Monitor Heart Rate Variability and Oxygen Saturation in Older People
Brief Title: Finger Wearable Device to Monitor Heart Rate Variability and Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2016.454
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Chronic obstructive airway disease (COPD) is common condition in old age and the perception of hypoxia is often impaired in some COPD patients. Therefor it is need to monitor oxygen saturation in older people with COPD. A finger wearable device has been developed to measure oxygen saturation and heart rate variability. The investigators therefore will perform a cross sectional study to evaluate the clinical application of this finger wearable device in the detection and management of COPD in older people.

Subject and method: 100 COPD subjects and 200 community dwelling older people without diagnosis of COPD will be recruited. Physical functioning and lung function test will be performed. Subjects will wear a finger wearable device to monitor heart rate variability and oxygen saturation and wear another wrist wearable device (Actigraph) to monitor physical activity and sleep for 6 days at the same time.

Statistical analysis: Statistical analysis will be made to examine the potential association between oxygen saturation and physical activity and sleep, and the association between heart rate variability and physical activity and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years old or more with or without COPD

Exclusion Criteria:

* Current smokers

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 COPD and 200 healthy older people
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
COPD | 6 days
  COPD as defined by lung function

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Hong Kong, Hong Kong